CLINICAL TRIAL: NCT00137280
Title: Implementing Effective, Collaborative Care for Schizophrenia
Brief Title: Implementing Effective, Collaborative Care for Schizophrenia (EQUIP-2)
Acronym: EQUIP-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: University of California, Los Angeles (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: Single | Purpose: Health Services Research
Other Study IDs: MNT 03-213; P30MH082760 (NIH)
Record Dates: First submitted 2005-08-25; First posted 2005-08-29 (Estimated); Results first posted 2014-10-15 (Estimated); Last update posted 2018-02-22 (Actual); Status verified 2018-01

CONDITIONS: Schizophrenia; Chronic Illness; Weight Gain; Psychotic Disorder
Keywords: Randomized Controlled Trial; Quality of Health Care; Health Services Research; Guidelines; Medical Informatics Computing; Services, Mental Health; Medicine, Evidenced-Based; Quality Assurance, Healthcare; Quality Indicators, Health Care; Veterans; Unemployment; Obesity; Quality Improvement
MeSH Terms: conditions — Schizophrenia; Chronic Disease; Weight Gain; Psychotic Disorders; Psychological Well-Being; Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: research assessors had minimal contact with staff involved in implementation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Collaborative Chronic Illness Care Model (Experimental): Collaborative Chronic Illness Care Model: A care model that integrates greater availability of clinical information, reorganizes the practice system and provider roles, fosters care coordination, and focuses on evidence-based protocols--specifically supported employment and wellness services for individuals with schizophrenia.
  Interventions: Behavioral: Collaborative Chronic Illness Care Model
- Usual Care (No Intervention): Usual Care

INTERVENTIONS:
Behavioral: Collaborative Chronic Illness Care Model — A care model that integrates greater availability of clinical information, reorganizes the practice system and provider roles, fosters care coordination, and focuses on evidence-based protocols--specifically supported employment and wellness services for individuals with schizophrenia.
  Arms: Collaborative Chronic Illness Care Model

SUMMARY:
This project evaluates the implementation and effectiveness of a care model to improve treatment for schizophrenia within the context of diverse VA practices and priorities. The project provides information to VA clinicians and managers about Veterans with schizophrenia or schizoaffective disorder who are overweight and/or who would like to return to competitive work. The project facilitates reorganization of care practices in order to get veterans needed and desired services around wellness and work. The project creates a platform that other clinical and research interventions can build upon to improve care, and is designed to inform a national strategy for implementing evidence-based care in schizophrenia.

DETAILED DESCRIPTION:
Objectives:

EQUIP-2 is a clinic-level controlled trial. From the four participating Veterans Integrated Services Networks (VISNs), eight specialty mental health programs were enrolled and assigned to care as usual or to receive an intervention supporting evidence-based quality improvement and use of a chronic illness care model. Participants are VISN 3 (James J. Peters VA; Northport VA); VISN 16 (Houston VA; Shreveport VA); VISN 17 (Waco VA; Temple VA); and VISN 22 (Long Beach VA; Greater Los Angeles VA). The objectives of this VA Quality Enhancement Research Initiative (QUERI) Service Directed Project are 1) assist in identifying and making available recovery-oriented services to veterans with schizophrenia; 2) implement information systems that efficiently and accurately identify patient status and who would be appropriate for these services; 3) implement a care model to support recovery-oriented care delivery; 4) evaluate, in a controlled trial, the effect of implementation on treatment delivery and patient outcomes; and 5) identify facilitators and barriers to wellness program participation in an effort to strengthen the weight management services available to patients with schizophrenia. The project studies intervention feasibility, acceptability, and impact on outcomes; performs qualitative analyses examining processes and variation in care model implementation and impact. Research includes a controlled trial of the impact of implementation, relative to usual care, on treatment quality. Participants include clinic staff and patients with schizophrenia. Data sources include interviews with participants, focus groups with a sub-set of patients, implementation documentation, the project informatics system, and VistA.

Methods:

The care model targets two clinical domains selected by the VISNs from the following: Supported Employment (SE), caregiver support, wellness programs, or clozapine. All 4 VISNs chose the same two targets: SE and wellness. The care model includes: 1) at each visit, routine collection of patient outcomes data and provision of decision support using a self-assessment kiosk; 2) provision of "psychiatric vital signs" to patients and clinicians at the time of the clinical encounter via report that prints from the kiosk; 3) education and activation of both clinicians and patients around the clinical targets; 4) regular reports identifying patients appropriate for services associated with these targets; and 5) facilitation of problem-solving and evidence-based quality improvement addressing any barriers to utilization of these services.

To inform future wellness implementation, in-depth, semi-structured interviews are conducted with patients who participated in wellness groups ("participants"), and with patients who were referred (because they were overweight or obese) but did not participate ("non-participants"). Participants consist of all enrolled patients who attended the wellness program with special attention to those patients who completed at least half of the wellness program. Non-participants consist of patients who were referred to the wellness program but did not attend. Clinicians were interviewed specifically regarding wellness implementation.

ELIGIBILITY:
Inclusion Criteria:

Clinicians and Managers:

* Psychiatrists, Case Managers, Nurses, Supported Employment workers Nutritionists, Local Recovery Coordinators, and Quality Improvement experts working at one of the participating VA Medical Centers

Patients:

* At least 18 years old
* Diagnosis of Schizophrenia, Schizoaffective, or schizophreniform disorder
* At least 1 treatment visit with a clinician at the clinic during the 6 months prior to enrollment and then at least 1 treatment visit with a clinician at the clinic during the 5 months of enrollment.

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1067 (Actual)
Dates: Start 2007-06-13 (Actual); Primary Completion 2010-03-05 (Actual); Study Completion 2011-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Stehle Young, MD MSHS, Principal Investigator — VA Greater Los Angeles Healthcare System, West Los Angeles, CA
Locations (8):
- United States (8):
  - VA Long Beach Healthcare System, Long Beach, CA, Long Beach, California
  - VA Greater Los Angeles Healthcare System, West Los Angeles, CA, West Los Angeles, California
  - Overton Brooks VA Medical Center, Shreveport, LA, Shreveport, Louisiana
  - VA Southern Nevada Healthcare System, North Las Vegas, NV, Las Vegas, Nevada
  - Northport VA Medical Center, Northport, NY, Northport, New York
  - James J. Peters VA Medical Center, Bronx, NY, The Bronx, New York
  - Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas
  - Central Texas Veterans Health Care System, Temple, TX, Temple, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Young AS, Niv N, Cohen AN, Kessler C, McNagny K. The appropriateness of routine medication treatment for schizophrenia. Schizophr Bull. 2010 Jul;36(4):732-9. doi: 10.1093/schbul/sbn138. Epub 2008 Nov 7. PMID 18997159
- [Result] Brown AH, Cohen AN, Chinman MJ, Kessler C, Young AS. EQUIP: implementing chronic care principles and applying formative evaluation methods to improve care for schizophrenia: QUERI Series. Implement Sci. 2008 Feb 15;3:9. doi: 10.1186/1748-5908-3-9. PMID 18279505
- [Result] Hamilton AB, Cohen AN, Young AS. Organizational readiness in specialty mental health care. J Gen Intern Med. 2010 Jan;25 Suppl 1(Suppl 1):27-31. doi: 10.1007/s11606-009-1133-3. PMID 20077148
- [Result] Young AS, Niv N, Chinman M, Dixon L, Eisen SV, Fischer EP, Smith J, Valenstein M, Marder SR, Owen RR. Routine outcomes monitoring to support improving care for schizophrenia: report from the VA Mental Health QUERI. Community Ment Health J. 2011 Apr;47(2):123-35. doi: 10.1007/s10597-010-9328-y. Epub 2010 Jul 25. PMID 20658320
- [Result] Cohen AN, Chinman MJ, Hamilton AB, Whelan F, Young AS. Using patient-facing kiosks to support quality improvement at mental health clinics. Med Care. 2013 Mar;51(3 Suppl 1):S13-20. doi: 10.1097/MLR.0b013e31827da859. PMID 23407006
- [Result] Hamilton AB, Cohen AN, Glover DL, Whelan F, Chemerinski E, McNagny KP, Mullins D, Reist C, Schubert M, Young AS. Implementation of evidence-based employment services in specialty mental health. Health Serv Res. 2013 Dec;48(6 Pt 2):2224-44. doi: 10.1111/1475-6773.12115. Epub 2013 Oct 21. PMID 24138608
- [Result] Pedersen ER, Huang W, Cohen AN, Young AS. Alcohol use and service utilization among veterans in treatment for schizophrenia. Psychol Serv. 2018 Feb;15(1):21-30. doi: 10.1037/ser0000109. Epub 2017 Mar 13. PMID 28287773

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were selected randomly from the population of individuals with schizophrenia receiving care at VA mental health clinics. All clinicians and managers at mental health clinics were selected.
Pre-assignment Details: Patients were excluded if they did not meet inclusion criteria, refused to participate, or were not approached about participation. Staff were excluded if they refused to participate.
Groups:
- Usual Care: Continue with usual care
Period: Overall Study
Arm/Group | Collaborative Chronic Illness Care Model | Usual Care
Started | 389 | 412
Completed | 305 | 357
Not Completed | 84 | 55

BASELINE CHARACTERISTICS:
Population: People with schizophrenia
Groups:
- Total: Total of all reporting groups
Arm/Group | Collaborative Chronic Illness Care Model | Usual Care | Total
Number analyzed (Participants) | 389 | 412 | 801
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.0 (9.3) | 54.5 (9.5) | 54.3 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 39 | 69
  Male | 359 | 373 | 732
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 10 | 13
  Asian | 3 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 4 | 1 | 5
  Black or African American | 160 | 195 | 355
  White | 175 | 180 | 355
  More than one race | 11 | 4 | 15
  Unknown or Not Reported | 33 | 19 | 52
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 72 | 28 | 100
  Not Hispanic or Latino | 312 | 380 | 692
  Unknown or Not Reported | 5 | 4 | 9
Region of Enrollment [Number; unit: participants]
  United States | 389 | 412 | 801
Duration with Schizophrenia, years [Mean (Standard Deviation); unit: years] | 26.2 (11.7) | 25.8 (12.7) | 26.0 (12.3)
Psychotropic medications by weight gain potential [Number; unit: participants] — Participants are only counted in one category; Participants are counted in the highest weight gain potential category.
  participants
    High Weight Gain Potential | 70 | 65 | 135
    Moderate Weight Gain Potential | 149 | 158 | 307
    Low Weight Gain Potential | 96 | 92 | 188
    Unknown/Not Reported | 74 | 97 | 171
Weight, kilograms [Mean (Standard Deviation); unit: kilograms] | 94.6 (20.4) | 93.0 (20.1) | 93.8 (20.2)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 30.2 (6.1) | 29.9 (6.5) | 30.1 (6.3)
Diagnosis of Diabetes [Number; unit: participants]
  Yes | 120 | 118 | 238
  No | 269 | 294 | 563
Waist Circumference, centimeters [Mean (Standard Deviation); unit: centimeters] | 104.9 (16.3) | 104.3 (15.7) | 104.6 (16.0)
Psychotic Symptoms, Brief Psychiatric Rating Scale [Mean (Standard Deviation); unit: units on a scale] — The Brief Psychiatric Rating Scale includes a number of scales that measure domains of psychopathology. Item scores and scale scores range from 1 (none) to 7 (extremely severe). The psychotic symptoms scale measures severity of psychosis.
  units on a scale | 2.3 (1.3) | 2.5 (1.3) | 2.4 (1.3)
Negative Symptoms, Brief Psychiatric Rating Scale [Mean (Standard Deviation); unit: units on a scale] — The Brief Psychiatric Rating Scale includes a number of scales that measure domains of psychopathology. Item scores and scale scores range from 1 (none) to 7 (extremely severe). The negative symptoms scale measures severity of negative symptoms.
  units on a scale | 1.5 (0.8) | 2.0 (1.3) | 1.8 (0.8)
Functioning, Global Assessment of Functioning Scale [Mean (Standard Deviation); unit: units on a scale] — The Global Assessment of Functioning Scale consists of three scales: occupational functioning, social functioning, and symptomatic functioning. Each scale ranges from 1 (worst possible functioning) to 100 (superior functioning).
  units on a scale
    Occupational Functioning | 39.5 (20.6) | 38.2 (16.8) | 38.8 (18.8)
    Social Functioning | 53.4 (14.1) | 54.4 (12.9) | 53.9 (13.5)
    Symptomatic Functioning | 53.4 (15.1) | 50.2 (13.8) | 51.7 (14.5)

OUTCOME MEASURES:

1. Primary Outcome: The Effect of Care Model Implementation on Treatment Appropriateness: Weight Service Utilization
Description: The number of participants with one or more weight service appointments in the one year during implementation (implementation sites versus control sites) for those participants who were overweight at the baseline interview (e.g., eligible for weight services). This only includes participants who were overweight at the baseline interview (e.g., eligible for weight services).
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | Collaborative Chronic Illness Care Model | Usual Care
Number analyzed (Participants) | 308 | 315
participants | 73 | 38
Statistical Analysis 1: Comparison: Collaborative Chronic Illness Care Model vs Usual Care; Test type: Superiority or Other; p < 0.01, Regression, Logistic; Odds Ratio (OR) = 2.3, 95% CI 2-sided [1.47 to 3.58] — Comparison group is the control (denominator)

2. Primary Outcome: The Effect of Care Model Implementation on Treatment Appropriateness: Patient Weight Outcomes
Description: Analysis of Covariance (ANCOVA) was used to examine weight gained during treatment in implementation versus control groups. The dependent variable was final weight. Baseline weight, weight 6 months prior to baseline, and baseline psychotic and negative symptom subscales were included as covariates. The inclusion of weight 6 months prior to baseline served to control for subjects' weight gain/loss trajectories prior to entering the study. The two-way interactions of group by covariates were also included in the model.
Time Frame: 1 year
Measure: Least Squares Mean (Standard Error); unit: pounds
Arm/Group | Collaborative Chronic Illness Care Model | Usual Care
Number analyzed (Participants) | 273 | 332
pounds | 208.1 (.92) | 207.2 (.83)
Statistical Analysis 1: Comparison: Collaborative Chronic Illness Care Model vs Usual Care; Test type: Superiority or Other; p = .03, ANCOVA; Mean Difference (Final Values) = 13.02, Standard Error of Mean 5.93

3. Primary Outcome: The Effect of Care Model Implementation on Treatment Appropriateness: Supported Employment Utilization
Description: The number of participants with one or more Supported Employment appointments in the one year during implementation (implementation sites versus control sites) for those participants who endorsed a desire to return to work at the baseline interview (e.g., eligible for Supported Employment services). This only includes participants who endorsed a desire to return to work at the baseline interview (e.g., eligible for Supported Employment services).
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | Collaborative Chronic Illness Care Model | Usual Care
Number analyzed (Participants) | 194 | 212
participants | 32 | 17
Statistical Analysis 1: Comparison: Collaborative Chronic Illness Care Model vs Usual Care; Test type: Superiority or Other; p < 0.01, Regression, Logistic; Odds Ratio (OR) = 2.3, 95% CI 2-sided [1.22 to 4.34] — Comparison group is the control (denominator)

4. Primary Outcome: The Effect of Care Model Implementation on Treatment Appropriateness: Patient Employment Outcomes
Description: Chi-square analysis was used to examine competitive employment gained during treatment in implementation versus control groups. The dependent variable was competitive employment. Individuals included were only those who expressed interest in returning to work at both the baseline and follow-up interview time-points.
Time Frame: 1 year
Measure: Number; unit: competitive employment
Arm/Group | Collaborative Chronic Illness Care Model | Usual Care
Number analyzed (Participants) | 96 | 148
competitive employment | 14 | 12
Statistical Analysis 1: Comparison: Collaborative Chronic Illness Care Model vs Usual Care; Test type: Superiority or Other; p = .11, Chi-squared

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Collaborative Chronic Illness Care Model | Usual Care
Serious Adverse Events (participants affected / at risk) | 0/389 | 0/412
Other Adverse Events (participants affected / at risk) | 0/389 | 0/412

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes